CLINICAL TRIAL: NCT02143596
Title: Neuroprotective Therapy and Therapeutic Target in Emergency Department
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100-4630C
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Stroke; Dehydration
Keywords: stroke; dehydration; prognosis
MeSH Terms: conditions — Stroke; Dehydration | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bun/Cr based hydration (Active Comparator): receive intravenous normal saline infusion and adjust infusion rate by Bun/Cr followed in the first 72 hours
  Interventions: Other: normal saline
- control (No Intervention): receive intravenous normal saline infusion as clinician's adjustment

INTERVENTIONS:
Other: normal saline — the infusion rate of normal saline is determinated by clinicians according to Bun/Cr ratio followed
  Arms: Bun/Cr based hydration

SUMMARY:
The investigators studied laboratory measurements and previously identified risk factors to identify factors predictors of early deterioration following stroke. A prospective observational study of 196 patients with first-time acute ischemic stroke was performed. Following multivariate analysis, only a Bun/Cr >15 was independent predictor of SIE. These patients were 3.41-fold more likely to have SIE (P=0.008). The elevated Bun/Cr ratio indicates relative dehydration of the patients. An immediate intervention for such patients should be the maintenance of proper hydration.

DETAILED DESCRIPTION:
In previous reports, many predictors of early deterioration after ischemic stroke have been proposed and studied, yet the results remain controversial. For example, several studies have been performed to ascertain whether cerebral or systemic causes are the major determinants of stroke deterioration. The findings, however, have been inconsistent. Measures of overall status and stroke severity (low initial Canadian Stroke Severity score, low initial National Institutes of Health Stroke Scale score, early CT findings of stroke severity, and changes in cerebral blood flow affecting the ischemic penumbra as measured by positron emission tomography and single photon emission computed tomography imaging have been shown to predict early deterioration. Laboratory tests for coagulation markers (fibrinogen, D-dimers), inflammatory markers (increased interleukin-6, decreased interleukin-10), serum glucose at admission, hematocrit and physiological parameters, such as blood pressure (both elevated and decreased), and body temperature have been identified as predictors of early deterioration. In addition, patient medical history (diabetes mellitus, atherosclerosis, chronic heart disease) has also been associated with early stroke deterioration. These differing findings may be due to variations in study design, patient populations, selection and exclusion criteria, and the criteria used for defining early deterioration.

A further complication in trying to determine predictors of early deterioration after stroke is that different stroke subtypes may manifest differently in terms of clinical changes before deterioration. In most of the aforementioned studies, no attempt was made to differentiate among stroke subtypes. While others have shown that some proposed markers are statistically significant only for certain stroke subtypes. A predictor of early deterioration that is equally applicable to all stroke subtypes is needed.

The investigators studied laboratory measurements and previously identified risk factors to identify factors predictors of early deterioration following stroke. A prospective observational study of 196 patients with first-time acute ischemic stroke was performed. Following multivariate analysis, only a Bun/Cr >15 was independent predictor of SIE. These patients were 3.41-fold more likely to have SIE (P=0.008). The elevated Bun/Cr ratio indicates relative dehydration of the patients.

Monitoring of hydration status would also appear to be critical in these patients. Being able to accurately identify patients at risk for early deterioration following stroke will allow for the design of clinical trials of stroke intervention targeting patients with SIE. The investigators need further tests to confirm if the maintenance of proper hydration improve outcome in patients with a Bun/Cr ratio higher than 15.

ELIGIBILITY:
Inclusion Criteria:

* acute stroke

Exclusion Criteria:

* 1.the time between the onset of neurological symptoms and emergency department presentation are more than 12 hours

  2.required fibrinolytic therapy

  3.required surgical intervention

  4.underline disease including congestive heart failure, chronic renal failure ( Cr>2 mg/dl) , liver cirrhosis, chronic obstructive pulmonary disease

  5. initial systolic blood pressure>200 or diastolic blood pressure > 120 mmHg

  6.initial systolic blood pressure<100 mmHg

  7.oxygen saturation less than 92% ( room air )

  8. require diuretics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2010-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
rate of stroke in evolution | 72 hours after admission

CONTACTS AND LOCATIONS:
Overall Officials: Leng C Lin, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Chiayi City, Taiwan

REFERENCES:
- [Background] Lin LC, Yang JT, Weng HH, Hsiao CT, Lai SL, Fann WC. Predictors of early clinical deterioration after acute ischemic stroke. Am J Emerg Med. 2011 Jul;29(6):577-81. doi: 10.1016/j.ajem.2009.12.019. Epub 2010 Apr 2. PMID 20825831
- [Background] Tei H, Uchiyama S, Ohara K, Kobayashi M, Uchiyama Y, Fukuzawa M. Deteriorating ischemic stroke in 4 clinical categories classified by the Oxfordshire Community Stroke Project. Stroke. 2000 Sep;31(9):2049-54. doi: 10.1161/01.str.31.9.2049. PMID 10978028